CLINICAL TRIAL: NCT02640651
Title: An Open Label Pilot Study of Transcranial Direct Current Stimulation in Adults With ADHD
Brief Title: An Study of Transcranial Direct Current Stimulation in Adults With ADHD
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of study staff
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Craig B. Surman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P001728
Record Dates: First submitted 2015-09-23; First posted 2015-12-29 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DC-Stimulator (PLUS version) (Experimental): For tDCS stimulation, anodal stimulation of the right dorsolateral prefrontal cortex will be performed for twenty minutes at 2mA. The current will be applied by a battery-driven tDCS stimulator via a pair of saline-soaked sponge electrodes (25 cm2 surface). The anodal electrode will be placed on the scalp at the F4 position according to the international 10-20 EEG coordinate system. 20 minute tDCS sessions will be conducted ten times over a two week period
  Interventions: Device: DC-Stimulator (PLUS version)

INTERVENTIONS:
Device: DC-Stimulator (PLUS version) — transcranial direct current stimulation

SUMMARY:
The purpose of this pilot study is to determine whether transcranial direct current stimulation safely and effectively improves symptoms of ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults 18-65 years of age.
* A diagnosis of childhood onset ADHD, meeting the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) [American Psychiatric Association, 2013] criteria, including at least 5 moderate inattentive or impulsive-hyperactive symptoms, and onset of several symptoms of inattentive or of impulsive/hyperactive traits by the age of 12.
* English-speaking.

Exclusion Criteria:

- Current or past history of mental retardation, severe sensory impairment such as deafness or blindness, hypomania, mania, psychosis, suicidal or homicidal behavior.

Current moderate to severe symptoms of a mental health condition other than ADHD, assessed using a clinical evaluation and the Adult Self Report Scale that, in the judgment of the investigator, may jeopardize subject safety or interfere with their ability to participate in the study. Specifically, this will include current clinical diagnosis of moderate to severe major depression, or a score on the depressive problem subscale of the ASRS that falls in the clinically significant range.

* Substance use disorder within the past 6 months.
* Any significant medical condition, that, in the judgment of the investigator, may jeopardize subject safety.
* Pregnant females.
* Inability or unwillingness to participate in study procedures.
* Contraindication to tDCS: history of epilepsy, metallic implants in the head and neck, brain stimulators, vagus nerve stimulators, VP shunt, or pacemakers.
* Skin conditions that may make the application of, treatment with, and removal of the tDCS hardware painful as per the discretion of the clinician.
* Current use of a medication considered to be therapeutic for ADHD. If a subject is taking a medication that is considered by study investigators to potentially treat ADHD (eg. a stimulant, atomoxetine, buproprion, modafanil, serotonin-norepinephrine reuptake inhibitor, guanfacine or clonidine) they must stop use of this medication for at least 5 half lives of the drug under physician guidance prior to study participation. Subjects will not enter the study if it would require stopping a medication that is optimally and comfortably managing a clinical concern.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Adult ADHD Investigator Symptom Rating Scale (AISRS) | Baseline to 2 weeks
  Each of the individual DSM-V symptoms of ADHD is rated 0 to 3 on a scale of severity.
Behavior Rating Inventory of Executive Function-Adult (BRIEF-A) | Baseline to 2 weeks
  Assesses levels of executive function deficits
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline to 2 weeks
  A computer-based system designed to assess executive functioning

CONTACTS AND LOCATIONS:
Overall Officials: Craig Surman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States